CLINICAL TRIAL: NCT00806403
Title: Very Early Initiation of Treatment With Thrombolysis and Low Molecular Weight Heparin, Versus Abciximab and Low Molecular Weight Heparin Followed by Percutaneous Coronary Intervention, for Acute ST-Elevation Myocardial Infarction
Brief Title: Comparison Between Thrombolysis and Primary Percutaneous Coronary Intervention (PCI) to Treat ST-Segment Elevation Myocardial Infarction
Acronym: SWEDES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Stockholm South General Hospital (Other); Region Örebro County (Other); Norra Alvsborgs Lans Hospital, Trollhattan (Unknown); Varberg Hospital, Sweden (Other)
Responsible Party: Lars Grip, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWEDES 23/09/01
Record Dates: First submitted 2008-11-07; First posted 2008-12-10 (Estimated); Results first posted 2008-12-10 (Estimated); Last update posted 2008-12-10 (Estimated); Status verified 2008-11

CONDITIONS: Acute Myocardial Infarction
Keywords: thrombolysis; primary PCI; abciximab; ST-segment resolution; TIMI flow
MeSH Terms: interventions — reteplase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- thrombolysis (Active Comparator)
  Interventions: Drug: reteplase 10+10 U
- invasive (Active Comparator)
  Interventions: Procedure: primary PCI

INTERVENTIONS:
Drug: reteplase 10+10 U — comparison to primary PCI
  Other Names: Rapilysin
  Arms: thrombolysis
Procedure: primary PCI — comparison to thrombolysis
  Other Names: primary percutaneous coronary intervention
  Arms: invasive

SUMMARY:
The main objective is to compare a fibrinolytic strategy with an interventional strategy initiated as early as possible, preferably in the pre-hospital phase, with respect to resolution of ST-segment elevation at 120 minutes after inclusion and Thrombolysis In Myocardial Infarction (TIMI) flow grade evaluated at a mandated coronary angiography 5 to 7 days after inclusion.

DETAILED DESCRIPTION:
Patients in the fibrinolytic group received an intravenous injection of 30 mg enoxaparin followed by subcutaneous injections of 1 mg/kg body weight every 12 hours during hospital stay.

Patients in the invasive group were given an intravenous injection of enoxaparin of (0.75 mg/kg body weight) and abciximab as a intravenous bolus (0.25 mg/kg body weight) followed by a 12 hour infusion (10 microg/minute).

Secondary outcome measures were death, myocardial infarction and stroke alone or as a composite at 30 days.

Data on use of health care resources, loss of production and health-related quality of life were collected during one year. Cost-effectiveness was determined by comparing costs and quality-adjusted survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting within 6 h after onset of chest pain lasting for more than 30 min and with significant ST-segment elevation on ECG.

Exclusion Criteria:

* BP >180/110
* Known bleeding disorder
* Cardiogenic shock
* CPR>10 min
* Ongoing anticoagulant therapy
* Renal insufficiency
* Weight >120 kg

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2001-11; Primary Completion 2003-06 (Actual); Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Grip, M.D. PhD, Principal Investigator — Sahlgren's University Hospital/S; Leif Svensson, M.D. PhD, Study Chair — Stockholm South General Hospital; Johan Herlitz, M.D. PhD, Study Chair — Sahlgren's University Hospital/S; Mikael Dellborg, M.D. PhD, Study Chair — Sahlgren's University Hospital/O; Ake Ohlsson, M.D. PhD, Study Chair — Stockholm South General Hospital; Mikael Aasa, M.D., Study Chair — Stockholm South General Hospital
Locations (5):
- Sweden (5):
  - Sahlgrenska University Hospital, Gothenburg
  - Orebro University Hospital, Örebro
  - Sodersjukhuset, Stockholm
  - Norra Alvsborgs lans Hospital, Trollhättan
  - Varberg Hospital, Varberg

REFERENCES:
- [Result] Svensson L, Aasa M, Dellborg M, Gibson CM, Kirtane A, Herlitz J, Ohlsson A, Karlsson T, Grip L. Comparison of very early treatment with either fibrinolysis or percutaneous coronary intervention facilitated with abciximab with respect to ST recovery and infarct-related artery epicardial flow in patients with acute ST-segment elevation myocardial infarction: the Swedish Early Decision (SWEDES) reperfusion trial. Am Heart J. 2006 Apr;151(4):798.e1-7. doi: 10.1016/j.ahj.2005.09.013. PMID 16569536
- [Result] Aasa M, Kirtane AJ, Dellborg M, Gibson MC, Prahl-Abrahamsson U, Svensson L, Grip L. Temporal changes in TIMI myocardial perfusion grade in relation to epicardial flow, ST-resolution and left ventricular function after primary percutaneous coronary intervention. Coron Artery Dis. 2007 Nov;18(7):513-8. doi: 10.1097/MCA.0b013e3282c1fdb6. PMID 17925603
- [Derived] Aasa M, Henriksson M, Dellborg M, Grip L, Herlitz J, Levin LA, Svensson L, Janzon M. Cost and health outcome of primary percutaneous coronary intervention versus thrombolysis in acute ST-segment elevation myocardial infarction-Results of the Swedish Early Decision reperfusion Study (SWEDES) trial. Am Heart J. 2010 Aug;160(2):322-8. doi: 10.1016/j.ahj.2010.05.008. PMID 20691839

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From Nov. 2001 to May 2003. Cardiology Departments
Groups:
- Thrombolysis: Reteplase 10U+10U i v plus enoxaparin 30 mg i v at first contact (prehospitally or in hospital) followed by enxaparin 1 mg/kg bodyweight s c every 12 h during hospital stay.
- Invasive: 500 mg aspirin p o and enoxaparin 0,75 mg/kg bodyweight plus a bolus of abciximab o,25 mg/kg bodyweight i v at first contact (prehospitally or in hospital). Therafter immediate transport to a catheterization lab for PCI. A loading dose of Clopidogrel 300 mg was given to stented patients immediately after PCI and continued for 3 months. Abciximab was given as an infusion of 10 mikrog/min for 12 h.
Period: Overall Study
Arm/Group | Thrombolysis | Invasive
Started | 104 | 101
Completed | 100 | 98
Not Completed | 4 | 3
Not completed — Death | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Thrombolysis | Invasive | Total
Number analyzed (Participants) | 104 | 101 | 205
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 55 | 49 | 104
  >=65 years | 49 | 52 | 101
Age Continuous [Mean (Standard Deviation); unit: years] | 64.3 (12.4) | 65.3 (10.9) | 64.8 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 27 | 53
  Male | 78 | 74 | 152
Region of Enrollment [Number; unit: participants]
  Sweden | 104 | 101 | 205

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With ST-segment Elevation Resolution Equal or More Than 50%
Description: ST-segment elevation resolution was measured in the lead with most prominent ST elevation at time of inclusion
Time Frame: 120 minutes after inclusion
Population: Analysis was made on intention to treat(ITT) basis.Patients with electrocardiograms (ECGs) suitable for analysis at inclusion and at 120 minutes therafter were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Thrombolysis | Invasive
Number analyzed (Participants) | 75 | 74
participants | 47 | 51
Statistical Analysis 1: Comparison: Thrombolysis vs Invasive; Null hypothesis:there is no difference in ST resolution at 120 minutes after inclusion between thrombolysis and primary PCI. The power calculation was based on the aim to prove a 50% reduction of failure to achive at least a 50% ST resolution (40% failure in thrombolysis group and 20% failure in Primary PCI group). With a power of 80% and a significance level of 0.05 (2-sided test), a total of 166 patients would be required; Test type: Superiority or Other; p = 0.56, Fisher Exact

2. Secondary Outcome: Death
Time Frame: 30 days
Population: Analysis was made on intention to treat (ITT) basis.
Measure: Number; unit: participants
Arm/Group | Thrombolysis | Invasive
Number analyzed (Participants) | 104 | 101
participants | 4 | 3
Statistical Analysis 1: Comparison: Thrombolysis vs Invasive; Test type: Superiority or Other; p = 1.00, Fisher Exact

3. Primary Outcome: Number of Patients With Thrombolysis In Myocardial Infarction (TIMI) Flow Grade 3
Description: Thrombolysis In Myocardial Infarction (TIMI) flow grade in the infarct related artery 5-7 days after inclusion.
Time Frame: 5-7 days after inclusion
Population: Patient were analyzed on intention to treat (ITT) basis. The per protocol angiography on day 5-7 after inclusion was used for analysis of Thrombolysis In Myocardial Infarction (TIMI) flow grade in the infarct related coronary artery.
Measure: Number; unit: participants
Arm/Group | Thrombolysis | Invasive
Number analyzed (Participants) | 65 | 79
participants | 35 | 56
Statistical Analysis 1: Comparison: Thrombolysis vs Invasive; Null hypothesis:there is no difference in number of patients with TIMI 3 flow at 5-7 days after inclusion between thrombolysis and primary PCI. The power calculation was based on the aim to prove a 65% reduction of failure to achive TIMI 3 flow (30% failure in thrombolysis group and 10% failure in Primary PCI group). With a power of 90% and a significance level of 0.05 (2-sided test), a total of 180 patients would be required; Test type: Superiority or Other; p = 0.04, Fisher Exact

4. Secondary Outcome: Reinfarction
Time Frame: 30 days
Population: Analysis made on intention to treat (ITT) basis.
Measure: Number; unit: Participants
Arm/Group | Thrombolysis | Invasive
Number analyzed (Participants) | 104 | 101
Participants | 2 | 0
Statistical Analysis 1: Comparison: Thrombolysis vs Invasive; Test type: Superiority or Other; p = 0.50, Fisher Exact

5. Secondary Outcome: Stroke
Time Frame: 30 days
Population: Analysis made on intention to treat (ITT) basis.
Measure: Number; unit: Participants
Arm/Group | Thrombolysis | Invasive
Number analyzed (Participants) | 104 | 101
Participants | 3 | 0
Statistical Analysis 1: Comparison: Thrombolysis vs Invasive; Test type: Superiority or Other; p = 0.21, Fisher Exact

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No